CLINICAL TRIAL: NCT02261246
Title: Trunk Motor Control Performance Before and After Spinal Manipulation Treatment
Acronym: TMCSMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We no longer have the resources to complete enrollment
Sponsor: Michigan State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jacek Cholewicki, Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NCCAM U19 AT006057 Project 2; 5U19AT006057-02 (NIH)
Record Dates: First submitted 2014-09-19; First posted 2014-10-10 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate treatment (Experimental): This arm receives spinal manipulation treatment shortly after enrollment
  Interventions: Procedure: Spinal manipulation treatment
- Delayed treatment (Experimental): This arm receives spinal manipulation treatment approximately 4 weeks after enrollment
  Interventions: Procedure: Spinal manipulation treatment
- Healthy control (no low back pain) (No Intervention): In this arm, healthy controls are tested at baseline.

INTERVENTIONS:
Procedure: Spinal manipulation treatment — Up to 4 sessions of spinal manipulation treatment (once per week).
  Arms: Delayed treatment; Immediate treatment

SUMMARY:
The overall goal of this project is to develop sensitive and objective clinical research tools for the assessment of trunk motor control. In order to accomplish this goal, the investigators aim to quantify changes in trunk motor control before and after spinal manipulation treatment. The investigators hypothesize that trunk motor control will improve in the low back pain participants after 4-weeks of spinal manipulation treatment. Additionally, the investigators will compare position and force trunk motor control between healthy controls and low back pain patients. The investigators hypothesize that baseline tests of position and force trunk motor control will be better in healthy individuals than low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet all of the inclusion criteria to participate in the study. Below is a list of inclusion criteria for ALL participants:

* Age 21-65 years
* Independently ambulatory
* Able to speak and read English
* Able to understand study procedures and to comply with them for the entire length of the study.

Below is an additional list of inclusion criteria for low back pain participants:

* Willing to be randomized to either immediate or delayed treatment group.
* Musculoskeletal pain - primarily in the lumbar region
* Pain rating greater or equal to 3 out of 10 as indicated on the Numeric Rating Scale for Pain
* Back Disability greater or equal to 26% as indicated on the Oswestry Disability Index

Exclusion Criteria:

All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation. Exclusion criteria will be self-reported. However, during each treatment session, the physicians will be watching for clinical signs and symptoms not consistent with physical findings that are suggestive of the presence of any of the exclusion criteria. In such a case, further treatment will be discontinued and the subject will be excluded.

Below is a list of exclusion criteria for ALL participants:

* Inability or unwillingness of individual to give written informed consent.
* Physical therapy or any other form of manual medicine (e.g., Osteopathic Manipulative Medicine, Chiropractic Manipulation, etc.), acupuncture or spinal injections within one month prior to study enrollment
* Workers' compensation benefits in the past 3 months or ongoing medical legal issues
* Possibly pregnant
* Extreme obesity (BMI>36)
* Currently using electrical implants (e.g., cardiac pacemakers, drug delivery pumps, etc.)

History of:

* Spinal surgery
* Spinal fracture
* Spinal infection (e.g., osteomyelitis)
* Cancer

Unresolved symptoms from:

* Head trauma
* Inner ear infection with associated balance and coordination problems
* Orthostatic hypotension
* Uncontrolled hypertension
* Vestibular disorder (e.g. vertigo)

Current diagnosis of:

* Significant spinal deformity (e.g., scoliosis > 20 degrees, torticollis)
* Ankylosing spondylitis
* Spondylolisthesis grades III or IV
* Cauda equine syndrome
* Rheumatoid arthritis
* Osteoporosis
* Angina or congestive heart failure symptoms
* Active bleeding or infection in the back
* Blindness
* Seizures
* Neurologic disease (e.g., Parkinson's disease, multiple sclerosis, cerebral palsy, Alzheimer's disease, amyotrophic lateral sclerosis, stroke or transient ischemic attack in the past year, cervical dystonia)

Conditions recognized by a physician any time during the study:

* Significant or worsening signs of neurologic deficit
* Symptoms are not consistent with mechanical findings
* Other conditions impeding protocol implementation

Below is an additional exclusion criterion for healthy control participants:

• Based on the minimal clinically important difference of 2 points (Childs et al., 2005), "healthy controls" with 2 points or greater pain on NRS will not be eligible to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 4 and from week 4 to 8 in trunk position tracking accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be in a seated position during the position tracking task and will wear a chest harness with an attached position sensor. The angular position of the trunk will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by moving their trunk. Accuracy will be determined by taking the difference between the target position signal and the actual trunk position (measured in degrees with string potentiometers).
Change from baseline to week 4 and from week 4 to 8 in trunk force tracking accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be in a seated position and will be asked to generate force with their trunk against a fixed pad. The pad will be attached to a load cell that monitors how much force is being generated by their trunk. The force level will be displayed on a monitor 1 meter in front of the participants and they will be asked to follow a moving target by generating force with their trunk. Accuracy will be determined by taking the difference between target force signal and the actual trunk force (measured in Newtons with the load cell).
Change from baseline to week 4 and from week 4 to 8 in trunk position stabilization accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be sitting in a seat mounted to a robotic platform (Mikrolar Hexapod Robot) and will wear a chest harness with an attached position sensor. The robotic platform will provide an angular perturbation to the participant about the lumbar spine in the sagittal plane while the participant is asked to maintain (stabilize) their trunk position in the upright posture. Accuracy will be determined by measuring the amount of trunk displacement (measured in degrees with string potentiometers) during the perturbation trial.
Change from baseline to week 4 and from week 4 to 8 in trunk force stabilization accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be sitting in a seat mounted to a robotic platform (Mikrolar Hexapod Robot) and will be asked to generate force with their trunk against a fixed pad. The pad will be attached to a load cell that monitors how much force is being generated by their trunk. The robotic platform will provide an angular perturbation to the participant about the lumbar spine in the sagittal plane while the participant is asked to maintain (stabilize) a static force level (projected on a screen in front of them) with their trunk (10% of the average maximum trunk moment). Accuracy will be determined by measuring the difference between the target force level and the actual force level maintained (measured in Newtons with a load cell) during the perturbation trial.
Change from baseline to week 4 and from week 4 to 8 in push stabilization accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be standing and will be asked to generate push force while holding onto a bar (arms along the body, elbows flexed at 90º). The bar will be attached to a load cell that monitors how much force is being applied with the hands. The robotic platform will provide a linear movement (perturbation) of the bar in the horizontal plane while the participant is asked to maintain (stabilize) a static force level (projected on a screen in front of them) with their hands (10% of the average maximum trunk moment). Accuracy will be determined by measuring the difference between the target force level and the actual force level maintained (measured in Newtons with a load cell) during the perturbation trial.
Change from baseline to week 4 and from week 4 to 8 in pull stabilization accuracy | Change from baseline to week 4 and from week 4 to 8
  Participants will be standing and will be asked to generate pull force while holding onto a bar (arms along the body, elbows flexed at 90º). The bar will be attached to a load cell that monitors how much force is being applied with the hands. The robotic platform will provide a linear movement (perturbation) of the bar in the horizontal plane while the participant is asked to maintain (stabilize) a static force level (projected on a screen in front of them) with their hands (10% of the average maximum trunk moment). Accuracy will be determined by measuring the difference between the target force level and the actual force level maintained (measured in Newtons with a load cell) during the perturbation trial.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) | The expected average is weekly for this outcome measure until the end of week 8
  Assesses weekly changes in physical function, anxiety, depression, fatigue, sleep, satisfaction with social role, and pain with PROMIS-29 questionnaire.
Change in concomitant medication | The expected average is weekly for this outcome measure until the end of week 8
  Assesses weekly changes in the use of medication for treating neck pain, including the type of medication and the quantity of medication (i.e., number of pills) with a questionnaire.
Change in back-related disability | The expected average is weekly for this outcome measure until the end of week 8
  Assesses weekly changes in functional limitations related to back pain with the Modified Oswestry Disability questionnaire.
Change in fear avoidance behavior | The expected average is weekly for this outcome measure until the end of week 8
  Assesses weekly changes in fear avoidance behavior using the Fear Avoidance Belief questionnaire.
Treatment effectiveness belief | This outcome measure will be assessed at baseline
  Assesses the patient's belief in how effective the treatment will be prior to treatment using the Credibility Expectancy questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Norman P Reeves, PhD, Principal Investigator — Sumaq Life LLC; Jacek Cholewicki, PhD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - MSU Osteopathic Manual Medicine, East Lansing, Michigan
  - MSU Musculoskeletal Rehabilitation, Lansing, Michigan
  - Michigan State University Center for Orthopedic Research, Lansing, Michigan

REFERENCES:
- [Background] Reeves NP, Popovich JM Jr, Priess MC, Cholewicki J, Choi J, Radcliffe CJ. Reliability of assessing trunk motor control using position and force tracking and stabilization tasks. J Biomech. 2014 Jan 3;47(1):44-9. doi: 10.1016/j.jbiomech.2013.10.018. Epub 2013 Oct 22. PMID 24262851
- See also: Website for Michigan State University Center for Orthopedic Research — http://orthopedicresearch.msu.edu/
- See also: Website for the National Center for Complementary and Alternative Medicine (Sponsor) — http://nccam.nih.gov/